CLINICAL TRIAL: NCT00006311
Title: Anxiety and Vagal Control of the Heart in Coronary Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 919; R01HL060826 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2006-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Depression; Heart Diseases; Death, Sudden, Cardiac; Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Depression; Heart Diseases; Death, Sudden, Cardiac; Arrhythmias, Cardiac

SUMMARY:
To examine the role of reduced vagal control of heart rate in the increased risk of cardiac mortality associated with anxiety in a population with established coronary artery disease (CAD). A second objective is to determine whether the effects of anxiety are independent of the effects of depression.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease continues to be the leading cause of death in the United States, despite risk factor reduction and technological advances in treatment options. Prospective studies implicate chronic anxiety as an independent risk factor for fatal coronary heart disease. In particular, anxiety increases the risk of sudden cardiac death substantially.

DESIGN NARRATIVE:

Nine hundred and fifty CAD patients were recruited for this study from patients hospitalized for elective cardiac catheterization. Anxiety was measured by the Hospital Anxiety Scale, the Spielberger Trait Anxiety Inventory, and the Crown-Crisp Phobic Anxiety Scale. Symptoms of depression were measured by the Montgomery-Asberg Depression Rating Scale, the Hospital Depression Scale, and the Beck Depression Inventory. Vagal control of heart rate was determined using power spectral analysis to measure two indices of vagal control: baroreceptor-mediated vagal reflex cardiac control, and respiratory sinus arrhythmia. Patients were followed at 6 months, l year, 2 years, and 3 years postcatheterization, and cardiac mortality data were obtained, including non-sudden and sudden cardiac death. The data generated by this study were used to examine the involvement of impaired vagal cardiac control in the risk of fatal coronary heart disease and sudden cardiac death associated with anxiety.

Specifically, the study examined: (1) the relationship between anxiety and cardiac mortality; (2) the relationship between anxiety and vagal control; (3) the role played by reduced vagal control in mediating anxiety-related risk; and (4) the relationship between depression, vagal control and cardiac risk. Findings of a relationship between anxiety, reduced vagal control and sudden cardiac death would suggest the potential importance of early intervention in cardiac patients with anxiety disorders and would underscore the benefit of aggressive monitoring of arrhythmias in this population, which may ultimately translate to reduced mortality rates.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-06; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Watkins — Duke University

REFERENCES:
- [Background] Watkins LL, Blumenthal JA, Carney RM. Association of anxiety with reduced baroreflex cardiac control in patients after acute myocardial infarction. Am Heart J. 2002 Mar;143(3):460-6. doi: 10.1067/mhj.2002.120404. PMID 11868052
- [Background] Hughes JW, Tomlinson A, Blumenthal JA, Davidson J, Sketch MH, Watkins LL. Social support and religiosity as coping strategies for anxiety in hospitalized cardiac patients. Ann Behav Med. 2004 Dec;28(3):179-85. doi: 10.1207/s15324796abm2803_6. PMID 15576256